CLINICAL TRIAL: NCT02228720
Title: The EXCEED Study: A Clinical Evaluation of the Drug-Eluting Propel Nova Sinus Implant When Placed in Peripheral Sinus Ostia to Maintain Patency
Brief Title: Clinical Evaluation of Propel Nova Sinus Implant in Peripheral Sinus Ostia
Acronym: EXCEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: P500-0414
Record Dates: First submitted 2014-06-25; First posted 2014-08-29 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-04

CONDITIONS: Chronic Sinusitis
Keywords: Chronic Sinusitis; Endoscopic Sinus Surgery

STUDY DESIGN:
Intervention Model Description: Propel Nova Sinus Implant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Propel Nova Sinus Implant (Experimental): Bioabsorbable, steroid-releasing sinus implant with 370 mcg of mometasone furoate released over 30 days
  Interventions: Device: Propel Nova Sinus Implant

INTERVENTIONS:
Device: Propel Nova Sinus Implant — Bioabsorbable, steroid-releasing sinus implant with 370 mcg of mometasone furoate released over 30 days
  Other Names: Propel Contour Sinus Implant (mometasone furoate, 370 mcg)

SUMMARY:
This is a feasibility study is to assess the performance, safety and initial signals of efficacy of the drug-eluting Propel Nova Sinus Implant when used in chronic sinusitis patients undergoing sinus surgery of peripheral sinus ostia.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm, open label feasibility study aiming to enroll at least 10 patients and a maximum of 15 patients to achieve 30 treated sinuses. The objective of this feasibility study is to assess the performance, safety and initial signals of efficacy of the drug-eluting Propel Nova Sinus Implant when used in chronic sinusitis (CS) patients undergoing sinus surgery of peripheral sinus ostia.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age.
* Patient is willing and able to comply with protocol requirements.
* Patient has CS as confirmed by CT scan and defined as symptoms lasting longer than 8 consecutive weeks in duration with inflammation of the mucosa of the nose and paranasal sinuses.
* Patient's condition and the planned intervention will involve at least two and a maximum of four peripheral sinuses (frontal or maxillary sinuses or combination of both).
* Patient is a candidate for a planned intervention involving sinus surgery in the operating room or office setting.
* Patient has nasal polyps no greater than grade 2.
* Patient with nasal polyps greater than 2 are eligible after their reduction/removal during ESS without significant complications that would confound the study results and leaving the patient's anatomy amenable to sinus implant placement, as judged by the operating physician.
* Female patients of child-bearing potential must not be pregnant and must agree to not become pregnant during the course of the study.
* Female patients of child-bearing potential must agree to use consistent and acceptable method/s of birth control during the course of the study.
* CS diagnosis confirmed and documented by CT Scan within 6 months of the procedure.
* Patient has a minimum total CT stage (Lund-Mackay method) of 6.
* Patient has disease in frontal and/or maxillary sinuses confirmed by CT scan.
* Planned ESS includes bilateral ethmoidectomy (if judged necessary), frontal sinus surgery using Draf II (A or B) dissection and/or balloon dilation, with minimum of 5-mm diameter opening created. In the case of maxillary sinus surgery, traditional antrostomy or balloon dilation, with or without removal of uncinate process, should be performed with minimum of 5-mm diameter opening created.
* Technique used for frontal or maxillary sinus surgery was the same on both sides (e.g. surgical dissection alone bilaterally, balloon dilation alone bilaterally, or both bilaterally)
* Septoplasty for access to the ostio-meatal complex is permitted.

Exclusion Criteria:

* Patient has presence of grade 3 or 4 polyposis, unless removed during surgery and preceding implant placement.
* Patient has presence of adhesions/scarring grades 3 or 4, unless removed during surgery and preceding implant placement.
* Patient has known history of immune deficiency (e.g., IGG subclass deficiency or IGA deficiency, HIV).
* Patient has concurrent condition requiring active chemotherapy and/or immunotherapy management for the disease (e.g., cancer, HIV, etc.).
* Patient has oral-steroid dependent condition such as COPD, asthma or other condition.
* Patient has known history of allergy or intolerance to corticosteroids or mometasone furoate.
* Patient has clinical evidence of acute bacterial sinusitis (e.g. acute increase in purulent discharge, fever, facial pain etc.).
* Patient has clinical evidence or suspicion of invasive fungal sinusitis (e.g. bone erosion on prior CT scan, necrotic sinus tissue, etc.).
* Patient has evidence of disease or condition expected to compromise survival or ability to complete follow-up assessments during the 90-day period.
* Patient is currently participating in another clinical trial.
* Patient has history of insulin dependent diabetes mellitus.
* Patient has previously undergone ESS and experienced a CSF leak or has residual compromised vision as a result of a complication in a prior ESS procedure.
* Patient has known dehiscence of the lamina papyracea.
* Patient has evidence of active viral illness (e.g., tuberculosis, ocular herpes simplex, chickenpox or measles).
* Significant complication during the current peripheral ostia surgery/such as excessive blood loss, CSF leak or punctured lamina papyracea.
* Current surgical intervention (operating room or office setting) is aborted for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Brown, MD, Principal Investigator — South Florida ENT Associates, PA
Locations (2):
- United States (2):
  - South Florida ENT Associates, Miami, Florida
  - Ohio Sinus Institute, Dublin, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Propel Nova Sinus Implant: Sinus stent with steroid coating (370 ug mometasone furoate)
  Propel Nova Sinus Implant: Sinus stent with steroid coating (370 ug mometasone furoate)
Period: Open Label - Baseline
Arm/Group | Propel Nova Sinus Implant
Started | 15
Completed | 15
Not Completed | 0
Period: Open Label - Day 30
Arm/Group | Propel Nova Sinus Implant
Started | 15
Completed | 14
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Open Label - Day 90
Arm/Group | Propel Nova Sinus Implant
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients and sinuses in whom placement of a Propel Nova Sinus Implant was attempted.
Groups:
- Propel Nova Sinus Implant: Steroid-releasing sinus implant with 370 mcg of mometasone furoate released over 30 days
Arm/Group | Propel Nova Sinus Implant
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.6 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13
Lund-Mackay Score (CT scan) [Mean (Standard Deviation); unit: units on a scale] — The severity of sinus mucosal inflammation or fluid accumulation scored as 0 (complete lucency), 1 (partial lucency) or 2 (complete opacity).
  units on a scale
    Frontal Sinuses | 2.5 (1.19)
    Maxillary Sinuses | 2.3 (0.98)

OUTCOME MEASURES:

1. Primary Outcome: Device Placement Success Rate
Description: Defined as successful access to and placement of the Propel Nova Sinus Implant in the frontal or maxillary sinus ostium within two attempts. Calculated as a proportion where the numerator is the number of successful device placements and the denominator is the number of attempted sinuses.
Time Frame: Baseline Procedure
Population: Attempted frontal and maxillary sinus ostia
Measure: Number; unit: Percentage of attempted sinuses
Units Other Than Participants: Sinuses
Groups:
- Propel Nova Sinus Implant: Bioabsorbable, steroid-releasing sinus implant with 370 mcg of mometasone furoate gradually released over time
Arm/Group | Propel Nova Sinus Implant
Number analyzed (Participants) | 15
Number analyzed (Sinuses) | 45
Percentage of attempted sinuses
  Frontal Sinuses: number analyzed (Sinuses) | 24
  Frontal Sinuses | 100
  Maxillary Sinuses: number analyzed (Sinuses) | 21
  Maxillary Sinuses | 95.2

2. Secondary Outcome: Ostial Patency
Description: Ostial patency grading scale from 0 (patent) to 1 (Occluded/Restenosed)
Time Frame: Baseline, Day 30, Day 90
Population: Frontal and maxillary sinus ostia
Measure: Number; unit: percentage of evaluable sinuses
Units Other Than Participants: Sinuses
Arm/Group | Propel Nova Sinus Implant
Number analyzed (Participants) | 15
Number analyzed (Sinuses) | 45
percentage of evaluable sinuses
  Baseline - Frontal Sinuses: number analyzed (Sinuses) | 24
  Baseline - Frontal Sinuses | 33.3
  Day 30 - Frontal Sinuses: number analyzed (Sinuses) | 22
  Day 30 - Frontal Sinuses | 100
  Day 90 - Frontal Sinuses: number analyzed (Sinuses) | 17
  Day 90 - Frontal Sinuses | 88.2
  Baseline - Maxillary Sinuses: number analyzed (Sinuses) | 21
  Baseline - Maxillary Sinuses | 57.1
  Day 30 - Maxillary Sinuses: number analyzed (Sinuses) | 21
  Day 30 - Maxillary Sinuses | 100
  Day 90 - Maxillary Sinuses: number analyzed (Sinuses) | 17
  Day 90 - Maxillary Sinuses | 94.1

3. Secondary Outcome: Adhesion/Scarring Grade 2 & 3
Description: Adhesion/scarring grading scale from 0 (No visible granulation/scarring), 1 (Minimal amount of scarring/contraction observed but non-obstructing the frontal or maxillary sinus ostium), 2 (moderate amount of obstructive scar tissue/contraction present in the frontal or maxillary sinus ostium), 3 (Significant scar tissue/ contraction causing obstruction of the frontal or maxillary sinus ostium)
Time Frame: Baseline, Day 30, Day 90
Population: Frontal and maxillary sinus ostia
Measure: Number; unit: percentage of evaluable sinuses
Units Other Than Participants: Sinuses
Arm/Group | Propel Nova Sinus Implant
Number analyzed (Participants) | 15
Number analyzed (Sinuses) | 45
percentage of evaluable sinuses
  Baseline - Frontal Sinuses: number analyzed (Sinuses) | 24
  Baseline - Frontal Sinuses | 33.4
  Day 30 - Frontal Sinuses: number analyzed (Sinuses) | 22
  Day 30 - Frontal Sinuses | 4.5
  Day 90 - Frontal Sinuses: number analyzed (Sinuses) | 17
  Day 90 - Frontal Sinuses | 11.8
  Baseline - Maxillary Sinuses: number analyzed (Sinuses) | 21
  Baseline - Maxillary Sinuses | 19.1
  Day 30 - Maxillary Sinuses: number analyzed (Sinuses) | 21
  Day 30 - Maxillary Sinuses | 0
  Day 90 - Maxillary Sinuses: number analyzed (Sinuses) | 19
  Day 90 - Maxillary Sinuses | 5.3

4. Secondary Outcome: Degree of Inflammation
Description: Inflammation visual analog scale (VAS) from 0 (no visible inflammation) to 100 (severe inflammation, involving significant and extensive erythema and edema and/or hypertrophy and/or polypoid changes)
Time Frame: Baseline, Day 30, Day 90
Population: Frontal and maxillary sinus ostia
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Sinuses
Arm/Group | Propel Nova Sinus Implant
Number analyzed (Participants) | 15
Number analyzed (Sinuses) | 45
units on a scale
  Baseline - Frontal Sinuses: number analyzed (Sinuses) | 24
  Baseline - Frontal Sinuses | 62.8 (23.14)
  Day 30 - Frontal Sinuses: number analyzed (Sinuses) | 22
  Day 30 - Frontal Sinuses | 28.1 (23.24)
  Day 90 - Frontal Sinuses: number analyzed (Sinuses) | 17
  Day 90 - Frontal Sinuses | 25.0 (25.23)
  Baseline - Maxillary Sinuses: number analyzed (Sinuses) | 21
  Baseline - Maxillary Sinuses | 51.6 (24.94)
  Day 30 - Maxillary Sinuses: number analyzed (Sinuses) | 21
  Day 30 - Maxillary Sinuses | 22.2 (13.55)
  Day 90 - Maxillary Sinuses: number analyzed (Sinuses) | 19
  Day 90 - Maxillary Sinuses | 14.1 (21.6)

5. Secondary Outcome: Sino-Nasal Outcome Test (SNOT) 22
Description: Validated, disease-specific, symptom-scoring instrument consisting of 22 questions, each scored by the patient on a scale of 0 (no problem) to 5 (problem as bad as it can be), resulting in a maximum total score of 110
Time Frame: Baseline, Day 30, Day 90
Population: Adult patients (≥ 18 years of age) diagnosed with chronic sinusitis with or without nasal/sinus polyposis who are candidates for endoscopic sinus surgery and in whom placement of the Propel Nova Sinus Implant is both feasible and medically appropriate
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Propel Nova Sinus Implant
Number analyzed (Participants) | 15
units on a scale
  Baseline | 42.6 (14.9)
  Day 30: number analyzed (Participants) | 14
  Day 30 | 21.5 (19.0)
  Day 90: number analyzed (Participants) | 14
  Day 90 | 20.6 (19.3)

ADVERSE EVENTS:
Time Frame: Day 90
Arm/Group | Propel Nova Sinus Implant
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 9/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propel Nova Sinus Implant (N=15)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propel Nova Sinus Implant (N=15)
Acute Sinusitis (Infections and infestations) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Vasovagal Reaction (General disorders) | 1 (1)
Sinus Drainage, green (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Crusting in nares (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No